CLINICAL TRIAL: NCT04739657
Title: Clinical Evaluation of A New High-speed and High-resolution Intravascular Ultrasound System: A Multi-center Prospective Control Study
Brief Title: Clinical Evaluation of A New High-speed and High-resolution Intravascular Ultrasound System
Acronym: NEW-IVUS
Status: Completed | Type: Observational
Sponsor: Insight Lifetech Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other); Guangdong Provincial People's Hospital (Other); Chinese PLA General Hospital (Other); Zhongda Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Other Study IDs: CTP-02-001
Record Dates: First submitted 2020-12-21; First posted 2021-02-04 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Percutaneous Coronary Intervention; Coronary Artery Disease; Chronic Total Occlusion of Coronary Artery; Left Main Coronary Artery Disease
Keywords: high-speed, high-resolution IVUS
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Subjects whose clinical conditions require stent implantation, and the interventional procedure of which needs the guidance of IVUS imaging.
  Interventions: Device: Insight Lifetech IVUS System; Device: Boston Scientific IVUS System

INTERVENTIONS:
Device: Insight Lifetech IVUS System — The Insight Lifetech IVUS System is intended for examination of coronary intravascular pathology only, including TrueVision IVUS diagnostic catheter and VivoHeart IVUS diagnostic device. IVUS imaging is used in patients who will undergo percutaneous coronary intervention.
  Other Names: IVUS diagnostic system
Device: Boston Scientific IVUS System — The Boston Scientific IVUS System is intended for the examination of coronary intravascular pathology only, including Opticross IVUS diagnostic catheter and iLAB IVUS diagnostic device. IVUS imaging is used in patients who will undergo percutaneous coronary intervention.
  Other Names: IVUS diagnostic system

SUMMARY:
Insight Lifetech Intravascular Ultrasound Diagnostic System (referred to as Insight Lifetech IVUS system below),is a new high-speed and high-resolution device for clearly defining vessel architecture and plaque morphology, providing quantitative and qualitative assessment of coronary arteries. Besides, IVUS has already an established role in guidance and optimization of percutaneous coronary intervention. This study will compare the differences, if any, between the intravascular ultrasound(IVUS) results measured by the two different IVUS diagnostic systems.

DETAILED DESCRIPTION:
Many studies have reported that IVUS is an accurate method for determining the size of the target vessel undergoing stent implantation , and the optimal stent deployment (complete stent expansion and apposition and lack of edge dissection or other complications after implantation). The novel 60 megahertz(60MHz) high-definition IVUS has evolved as a next-generation IVUS imaging technology to provide higher image resolution than conventional 40 megahertz(40MHz) IVUS but with sufficient imaging depth preserved for the assessment of the entire vessel wall structure.

Insight Lifetech IVUS system includes TrueVision IVUS diagnostic catheter and VivoHeart IVUS diagnostic console. It is a novel device with high speed, high resolution, and high image acquisition rate enabling high-speed pullback imaging up to 10mm/sec.

This study is a prospective, multi-center, randomized, single-blind, controlled study with the primary target of investigating the differences, if any, between IVUS measurement results by the Insight Lifetech IVUS system and Boston Scientific IVUS system, imaging catheter of which was available at 40MHz during the study. Other purposes included analyzing the feasibility of the Insight Lifetech IVUS system's high-speed pullback during the IVUS assessment. A total of 130 patients will be recruited from 5 centers in China.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 Years and older;
* Understand and willing to sign the informed consent form;
* Clinical evaluation shows that the coronary artery stent implantation and the intravascular ultrasound(IVUS) guidance is required.

Exclusion Criteria:

* Unable to understand or unwilling to sign the informed consent form;
* Clinically diagnosed with severe coronary artery spasms;
* Contraindicated to percutaneous coronary intervention (PCI);
* Presence of any other factor that the investigator deems is unsuitable for enrollment or completion of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease which needs the qualitative and quantitative assessment by IVUS mearsurement, for whom the IVUS guidance during pre- and post-PCI is required.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Mean Stent Area in square millimeter(MSA) | estimated 1 month on average, by a third-party corelab IVUS image post-analysis
  Comparison between the MSA measured by the Insight Lifetech Intravascular Ultrasound Diagnositic System and Boston Scientific Intravascular Ultrasound Diagnostic System, including mean relative deviation, confidence interval and standard deviation, as assessed by Bland-Altman analysis and Pearson correlation analysis.

SECONDARY OUTCOMES:
Clear Stent Length in millimeter (CSL) | estimated 1 month on average, by a third-party corelab IVUS image post-analysis
  Comparison between the CSL measured by the Insight Lifetech Intravascular Ultrasound Diagnostic System and Boston Scientific Intravascular Ultrasound Diagnostic System, including mean relative deviation, confidence interval and standard deviation, as assessed by Bland-Altman analysis and Pearson analysis.
Minimal Lumen Area in square millimeter(MLA) | estimated 1 month on average, by a third-party corelab IVUS image post-analysis
  Comparison between the MLA measured by the Insight Lifetech Intravascular Ultrasound Diagnostic System and Boston Scientific Intravascular Ultrasound Diagnostic System, including mean relative deviation, confidence interval and standard deviation, as assessed by Bland-Altman analysis and Pearson analysis.
The rate of detected stent malapposition, tissue prolapse and dissection | estimated 1 month on average, by a third-party corelab IVUS image post-analysis
  Detection rate of poor adherence, tissue prolapse and intercalation, for each system individually, and comparison between the two systems.
Stability of system (questionnaire) | estimated 1week on average, by opeartor's rating on questionaire
  Evaluate the stability of both systems concluded from all enrolled case using questionnaire, including below measures :
  1. the stability of IVUS examination ;
  2. the usability of system operation;
  3. the definition of images.
  For each system in 1., 2., and 3., only one of the following five ratings is given:
  * very stable/convenient/clear images;
  * stable/convenient/clear images, inspection was unaffected;
  * slightly unstable/inconvenient/unclear images, inspection was unaffected;
  * unstable/inconvenient/unclear images, inspection was affected; (in the order of 1./2./3.)
  * N/A.
  and is counted as 1 point for that particular rating. The distribution of the points in rating and how many points each rating individually owns are compared between the systems.
Maneuvering performance of catheter (questionnaire) | estimated 1week on average, by opeartor's rating on questionaire
  Evaluate the maneuvering performance of catheters in the two systems concluded from all enrolled case, including below measures :
  1. the pushability
  2. the crossability
  3. the angiographic visibility
  For each system in 1., 2., and 3., only one of the following five ratings is given:
  * excellent pushability/lesion crossability/visibility;
  * pushing met slight resistance/crossed lesion smoothly/good visibility, inspection was unaffected;
  * pushing met obvious resistance/crossed lesion after attempts/mediocre visibility, inspection was unaffected;
  * too resistant to push/unable to cross lesion/very poor visibility, inspection was affected; (in the order of 1./2./3.)
  * N/A.
  and is counted as 1 point for that particular rating. The distribution of the points in rating and how many points each rating individually owns are compared between the systems.
Device success rate | estimated 1day on average, by intraoperative monitoring
  Device success rate, defined as a valid IVUS image for each system, and comparison between the two systems.
Rate of device-related adverse effects | estimated 1day on average, by intraoperative monitoring
  Rate of device-related adverse effects, for each system individually, and comparison between the two systems.
Rate of thrombosis, diffuse lesion and re-stenosis as discerned by IVUS | estimated 1 month on average, by a third-party corelab IVUS image post-analysis
  Rate of thrombosis, diffuse lesion and re-stenosis discerned by each system individually, and comparison between the two systems.
Rate of plaque rupture and plaque properties as discerned by IVUS | estimated 1 month on average, by a third-party corelab IVUS image post-analysis
  Rates of plaque rupture, lipid-rich plaque, fibrous plaque and calcified plaque, discerned by each system individually, and comparison between the two systems.

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, MD, PhD, Principal Investigator — Zhongshan Hospital of Fudan Unviersity
Locations (5):
- China (5):
  - The General Hospital of the People's Liberation Army, Beijing
  - Guangdong Provincial People's Hospital, Guangzhou
  - Zhongda Hospital of Southeast University, Nanjing
  - Shanghai Zhongshan Hospital, Shanhai
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

REFERENCES:
- [Background] Li C, Yang J, Wang X, et al. CLINICAL VALIDATION OF A NEW INTRAVASCULAR ULTRASOUND SYSTEM: A COMPARATIVE ANALYSIS ON LENGTH MEASUREMENTS. J Am Coll Cardiol. 2022 Mar, 79 (9_Supplement) 827.